CLINICAL TRIAL: NCT01262651
Title: A Double Blind, Randomized, Placebo-controlled, Parallel Group Study of Sativex Oromucosal Spray (Sativex®; Nabiximols) as Adjunctive Therapy in Relieving Uncontrolled Persistent Chronic Pain in Patients With Advanced Cancer, Who Experience Inadequate Analgesia During Optimized Chronic Opioid Therapy
Brief Title: Sativex® for Relieving Persistent Pain in Participants With Advanced Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GW Pharmaceuticals Ltd (Industry)
Collaborators: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Organization: GWPharm (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GWCA0958; 2009-016064-36 (EudraCT Number)
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Pain; Advanced Cancer
Keywords: Cancer pain; Opioid therapy; Inadequate analgesia; Optimized chronic opioid therapy
MeSH Terms: conditions — Pain; Cancer Pain | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nabiximols (Experimental): Nabiximols was self-administered by participants as a 100 microliter (μL) oromucosal spray in the morning and evening, up to a maximum of 10 sprays per day for 5 weeks. Nabiximols oromucosal spray contained delta-9-tetrahydrocannabinol (THC) (27 milligram [mg]/milliliter [mL]):cannabidiol (CBD) (25 mg/mL), in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavoring. Each 100 μL actuation delivered 2.7 mg THC and 2.5 mg CBD.
  Interventions: Drug: Nabiximols
- Placebo (GA-0034) (Placebo Comparator): Placebo Comparator: Placebo (GA-0034) Placebo was self-administered by participants as a 100 μL oromucosal spray in the morning and evening, up to a maximum of 10 sprays per day for 5 weeks. Placebo oromucosal spray contained ethanol: propylene glycol (50:50)
  Interventions: Drug: Placebo (GA-0034)

INTERVENTIONS:
Drug: Nabiximols
  Other Names: Sativex®
  Arms: Nabiximols
Drug: Placebo (GA-0034)
  Arms: Placebo (GA-0034)

SUMMARY:
This 9-week study aimed to determine the efficacy, safety and tolerability of nabiximols (Sativex®) as an adjunctive treatment, compared with placebo in relieving uncontrolled persistent chronic pain in participants with advanced cancer.

Eligible participants were not required to stop any of their current treatments or medications.

DETAILED DESCRIPTION:
This 9-week, multi-center, double-blind, randomized, placebo-controlled study aimed to determine the efficacy, safety and tolerability of nabiximols, administered as an adjunctive treatment for 5 weeks, versus placebo. Eligible participants had advanced cancer, with a clinical diagnosis of cancer related pain which was not wholly alleviated by their current optimized opioid treatment.

Qualifying participants entered the study at screening and commenced a 5 to 14 day eligibility period. During this period, eligible participants had 3 consecutive days where pain severity remained within defined parameters, break-through opioid usage had not exceeded an average of 4 episodes per day, and maintenance opioid medication and dose had not changed. Eligible participants returned for randomization on Day 1 and were randomized to either the nabiximols or placebo treatment arm using a 1:1 allocation ratio. Participants began an initial titration period that lasted up to 14 days. The titration schedule required dosing to a minimum of 3 sprays per day, after which participants were allowed to individualize their dose (3 to 10 sprays per day) until Day 14 when that dose was then fixed for the remainder of the study. Participants returned at Day 22 and Day 36 (end of the randomized treatment period), or earlier if they terminated prematurely from the study. After the end of the 5-week treatment period, participants were offered the option of entering an open-label extension (OLE) study; a safety follow up visit (up to Day 43) was not required if the participant entered the OLE on Day 36. Participants who entered the OLE, up to 7 days after study completion had their follow-up assessments performed on the same day as their first OLE study visit. Participants that did not enter the OLE study had a safety follow up visit 14 days after treatment completion, which could be via telephone.

ELIGIBILITY:
Inclusion Criteria (abbreviated):

* The participant had advanced cancer for which there was no known curative therapy
* The participant had a clinical diagnosis of cancer related pain, which was not wholly alleviated with their current optimized opioid treatment
* The participant received an optimized maintenance dose of Step 3 opioid therapy, preferably with a sustained release preparation, but also allowing a regular maintenance dose of around the clock use of immediate release preparations
* The participant received a daily maintenance dose Step 3 opioid therapy of less than or equal to a total daily opioid dose of 500 mg/day of morphine equivalence (including maintenance and break-through opioids)
* The participant was using no more than one type of break-through opioid analgesia

Exclusion Criteria (abbreviated):

* The participant had any planned clinical interventions that would have affected their pain (for example, chemotherapy or radiation therapy where, in the clinical judgment of the investigator, these would be expected to affect pain)
* The participant was using or had used cannabis or cannabinoid-based medications within 30 days of study entry and is unwilling to abstain for the duration of the study
* The participant had experienced myocardial infarction or clinically significant cardiac dysfunction within the last 12 months or had a cardiac disorder that, in the opinion of the investigator, would have put the participant at risk of a clinically significant arrhythmia or myocardial infarction
* The participant had significantly impaired renal function
* The participant had significantly impaired hepatic function
* Female participants of child-bearing potential and male participants whose partner was of child-bearing potential, unless willing to ensure that they or their partner used effective contraception, for example, oral contraception, double barrier, intra-uterine device, during the study and for 3 months thereafter (however, a male condom was not to be used in conjunction with a female condom as this may not have proven effective)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2010-11-25 (Actual); Primary Completion 2015-07-02 (Actual); Study Completion 2015-07-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (68):
- United States (22):
  - Phoenix, Arizona
  - El Cajon, California
  - Gilroy, California
  - Brandon, Florida
  - Daytona Beach, Florida
  - Holiday, Florida
  - Jacksonville, Florida
  - Lynn Haven, Florida
  - Stuart, Florida
  - Winter Park, Florida
  - Newnan, Georgia
  - Stockbridge, Georgia
  - Shreveport, Louisiana
  - Saint Louis Park, Minnesota
  - Kansas City, Missouri
  - Berlin, New Jersey
  - Hendersonville, North Carolina
  - Winston-Salem, North Carolina
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Laredo, Texas
  - Salt Lake City, Utah
- Brussels, Belgium
- Bulgaria (3):
  - Gabrovo
  - Shumen
  - Varna
- Czechia (6):
  - České Budějovice
  - Hradec Králové
  - Most
  - Nová Ves pod Pleší
  - Ostrava-Poruba
  - Pilsen
- Germany (3):
  - Lünen
  - Stadtroda
  - Wetzlar
- Hungary (6):
  - Deszk
  - Kecskemét
  - Komárom
  - Miskolc
  - Nyíregyháza
  - Szekszárd
- Latvia (2):
  - Rēzekne
  - Riga
- Lithuania (3):
  - Klaipėda
  - Šiauliai
  - Vilnius
- Poland (5):
  - Bialystok
  - Bielsko-Biala
  - Gliwice
  - Poznan
  - Warsaw
- Puerto Rico (2):
  - Ponce
  - San Juan
- Romania (7):
  - Baia Mare
  - Brăila
  - Bucharest
  - Craiova
  - Oradea
  - Satu Mare
  - Suceava
- United Kingdom (8):
  - Bury
  - Bury St Edmunds
  - Edinburgh
  - Glasgow
  - Manchester
  - Norwich
  - Weston-super-Mare
  - Wolverhampton

REFERENCES:
- [Background] Lichtman AH, Lux EA, McQuade R, Rossetti S, Sanchez R, Sun W, Wright S, Kornyeyeva E, Fallon MT. Results of a Double-Blind, Randomized, Placebo-Controlled Study of Nabiximols Oromucosal Spray as an Adjunctive Therapy in Advanced Cancer Patients with Chronic Uncontrolled Pain. J Pain Symptom Manage. 2018 Feb;55(2):179-188.e1. doi: 10.1016/j.jpainsymman.2017.09.001. Epub 2017 Sep 18. PMID 28923526

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per the Statistical Analyses Plan, all randomized participants who received at least 1 dose of study drug were analyzed in the Intent-to-Treat (ITT) population as per randomized treatment group. However, if a participant randomized to placebo ever took a nabiximols dose, the participant was analyzed as nabiximols-treated in the Safety population.
Groups:
- Nabiximols: Nabiximols was self-administered by participants as a 100 microliter (μL) oromucosal spray in the morning and evening, up to a maximum of 10 sprays per day, for 5 weeks. Nabiximols oromucosal spray contained delta-9-tetrahydrocannabinol (THC) (27 milligram [mg]/milliliter [mL]):cannabidiol (CBD) (25 mg/mL), in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavoring. Each 100 μL actuation delivered 2.7 mg THC and 2.5 mg CBD.
- Placebo (GA-0034): Placebo was self-administered by participants as a 100 μL oromucosal spray in the morning and evening, up to a maximum of 10 sprays per day, for 5 weeks. Placebo oromucosal spray contained ethanol: propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavoring and colorings.
Period: Overall Study
Arm/Group | Nabiximols | Placebo (GA-0034)
Started | 199 | 198
Received at Least 1 Dose of Study Drug | 199 | 198
Safety Population | 199 | 198
ITT Population | 199 | 198
Completed | 141 | 150
Not Completed | 58 | 48
Not completed — Adverse Event | 40 | 35
Not completed — Withdrawal by Subject | 15 | 11
Not completed — Withdrawal by Investigator | 2 | 2
Not completed — Met Withdrawal Criteria | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one infusion of study drug.
Groups:
- Nabiximols: Nabiximols was self-administered by participants as a 100 μL oromucosal spray in the morning and evening, up to a maximum of 10 sprays per day, for 5 weeks. Nabiximols oromucosal spray contained THC (27 mg/mL):CBD (25 mg/mL), in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavoring. Each 100 μL actuation delivered 2.7 mg THC and 2.5 mg CBD.
- Total: Total of all reporting groups
Arm/Group | Nabiximols | Placebo (GA-0034) | Total
Number analyzed (Participants) | 199 | 198 | 397
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (12.0) | 60.7 (11.1) | 59.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 95 | 183
  Male | 111 | 103 | 214

OUTCOME MEASURES:

1. Primary Outcome: Percent Improvement From Baseline In Mean NRS Average Pain At End Of Treatment
Description: Participants indicated level of pain in the last 24 hours on an 11-point Numerical Rating Scale (NRS), where a score of 0 was "no pain" and 10 was "pain as bad as you can imagine". Baseline = mean score from first day of 3-day eligibility period through to the day before first dose of study drug. End of Treatment = mean score over last (up to) 7 days to the final pain score at End of Treatment or up until Day 35, whichever is earlier, or final score available (prematurely terminated).
  Percentage improvement from baseline (Imp%) was calculated as:
  Imp% = (Baseline pain NRS mean - End of Treatment pain NRS mean)/Baseline pain NRS mean * 100.
  For participants who died or withdrew due to disease progression, Imp% values were used. For participants who died or withdrew unrelated to disease progression before end of Week 5 (no diary data from Day 33 onwards), Imp% was zero for participants whose Imp% value was positive and it was Imp% for participants whose Imp% value was not positive.
Time Frame: Baseline, End of Treatment (Day 36)
Population: The ITT Population included all participants who were randomized, received at least 1 dose of study drug, and had at least 1 efficacy endpoint. Participants were analyzed according to the treatment group they were randomized to.
Measure: Median (Inter-Quartile Range); unit: percent improvement
Groups:
- Placebo (GA-0034): Placebo was self-administered by participants as a 100 μL oromucosal spray in the morning and evening, up to a maximum of 10 sprays per day, for 5 weeks. Placebo oromucosal spray contained ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavoring and colorings.
Arm/Group | Nabiximols | Placebo (GA-0034)
Number analyzed (Participants) | 199 | 198
percent improvement | 10.7 [0.0 to 30.0] | 4.5 [-2.9 to 25.7]
Statistical Analysis 1: Comparison: Nabiximols vs Placebo (GA-0034); Test type: Superiority; p = 0.0854, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 3.41, 95% CI 2-sided [0.00 to 8.16]

2. Secondary Outcome: Change From Baseline In Mean NRS Average Pain At End Of Treatment
Description: Participants indicated the level of pain experienced in the last 24 hours on an 11-point NRS, where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine." Change in mean NRS average pain was calculated as: End of Treatment NRS average pain score - Baseline NRS average pain score.
  A negative value indicates an improvement in average pain score from Baseline.
Time Frame: Baseline, End Of Treatment (Day 36)
Population: ITT Population included all participants who receive at least 1 dose of study drug, and had at least 1 efficacy endpoint. Participants were analyzed according to the treatment group they were randomized to.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nabiximols | Placebo (GA-0034)
Number analyzed (Participants) | 199 | 198
units on a scale | -0.8 (1.4) | -0.6 (1.5)

3. Secondary Outcome: Change From Baseline In Mean NRS Worst Pain At End Of Treatment
Description: Participants indicated the level of worst pain experienced in the last 24 hours on an 11-point NRS, where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine." Change in mean NRS worst pain was calculated as: End of Treatment NRS worst pain score - Baseline NRS worst pain score.
  A negative value indicates an improvement in worst pain score from Baseline.
Time Frame: Baseline, End of Treatment (Day 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nabiximols | Placebo (GA-0034)
Number analyzed (Participants) | 199 | 198
units on a scale | -0.9 (1.4) | -0.8 (1.6)

4. Secondary Outcome: Change From Baseline In Mean Sleep Disruption NRS At End Of Treatment
Description: Participants indicated the level of sleep disruption experienced in the last 24 hours on an 11-point NRS, where a score of 0 indicated "did not disrupt sleep" and a score of 10 indicated "completely disrupted (unable to sleep at all)." Change in mean sleep disruption NRS was calculated as: End of Treatment sleep disruption NRS score - Baseline sleep disruption NRS score.
  A negative value indicates an improvement in sleep disruption score from Baseline.
Time Frame: Baseline, End of Treatment (Day 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nabiximols | Placebo (GA-0034)
Number analyzed (Participants) | 199 | 198
units on a scale | -0.8 (1.7) | -0.5 (1.6)

5. Secondary Outcome: Subject Global Impression Of Change At Last Visit (Up To Day 36)
Description: The Subject Global Impression of Change (SGIC) was used to assess the overall status of the participant related to their cancer pain, with the markers "very much improved, much improved, slightly improved, no change, slightly worse, much worse, or very much worse". The SGIC was assessed at Day 36 or at which a participant's last evaluation was performed, such as in the case of early termination. Last visit refers to the last visit that a participant completed the assessment; this could be either Day 22 or Day 36.
Time Frame: Last Visit (up to Day 36)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nabiximols | Placebo (GA-0034)
Number analyzed (Participants) | 172 | 179
Participants
  Very Much Improved | 5 | 3
  Much Improved | 34 | 26
  Slightly Improved | 60 | 55
  No Change | 56 | 72
  Slightly Worse | 9 | 13
  Much Worse | 6 | 6
  Very Much Worse | 2 | 4

6. Secondary Outcome: Physician Global Impression Of Change At Last Visit (Up To Day 36)
Description: The Physician Global Impression of Change (PGIC) was used by the treating physician (investigator/sub-investigator) to assess if there was any change in the general functional abilities of the participant since prior to commencement of study medication, with the markers: "Very much worse, Much worse, Slightly worse, No change, Slightly improved, Much improved, Very much improved". Last visit refers to the last visit that a participant completed the assessment; this could be either Day 22 or Day 36.
Time Frame: Last Visit (up to Day 36)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nabiximols | Placebo (GA-0034)
Number analyzed (Participants) | 174 | 181
Participants
  Very much Improved | 6 | 3
  Much Improved | 37 | 25
  Slightly Improved | 56 | 50
  No Change | 41 | 75
  Slightly Worse | 25 | 19
  Much Worse | 7 | 5
  Very Much Worse | 2 | 4

7. Secondary Outcome: Patient Satisfaction Questionnaire At Last Visit (Up To Day 36)
Description: The Patient Satisfaction Questionnaire (PSQ) was used to assess level of satisfaction of the participant with the study drug, with the markers "Extremely satisfied, Very satisfied, Slightly satisfied, Neutral, Slightly dissatisfied, Very dissatisfied, Extremely dissatisfied". Last visit refers to the last visit that a participant completed the assessment; this could be either Day 22 or Day 36.
Time Frame: Last Visit (up to Day 36)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nabiximols | Placebo (GA-0034)
Number analyzed (Participants) | 171 | 179
Participants
  Extremely Satisfied | 7 | 3
  Very Satisfied | 42 | 38
  Slightly Satisfied | 42 | 37
  Neutral | 46 | 63
  Slightly Dissatisfied | 22 | 20
  Very Dissatisfied | 11 | 13
  Extremely Dissatisfied | 1 | 5

8. Secondary Outcome: Change From Baseline In Daily Total Opioid Use (Morphine Equivalent) At End Of Treatment
Description: The total daily opioid use (in morphine equivalence) was the sum of morphine equivalents of daily maintenance dose and break-through dose.
  Change in daily total opioid use was calculated as: End of Treatment daily total opioid use - Baseline daily total opioid use.
  A negative value indicates a decrease in use from Baseline.
Time Frame: Baseline, End of Treatment (Day 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg (morphine equivalent)
Arm/Group | Nabiximols | Placebo (GA-0034)
Number analyzed (Participants) | 199 | 198
mg (morphine equivalent) | 0.3 (34.7) | 0.6 (44.8)

9. Secondary Outcome: Change From Baseline In Daily Maintenance Opioid Dose (Morphine Equivalent) At End of Treatment
Description: The prescribed daily quantity of opioid maintenance dose was calculated as the product of dose per use and daily frequency of use. Participants were asked: "Have you used your maintenance dose painkiller today as prescribed?" If the participant answered "No" to the question, the daily opioid maintenance dose usage on that day was set to 0.
  Change in daily maintenance opioid dose was calculated as: End of Treatment daily maintenance opioid dose - Baseline daily maintenance opioid dose.
  A negative value indicates a decrease in dose from Baseline.
Time Frame: Baseline, End of Treatment (Day 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg (morphine equivalent)
Arm/Group | Nabiximols | Placebo (GA-0034)
Number analyzed (Participants) | 199 | 198
mg (morphine equivalent) | 0.2 (20.9) | -1.3 (38.7)

10. Secondary Outcome: Change From Baseline In Daily Break-through Opioid Dose (Morphine Equivalent) At End Of Treatment
Description: Daily break-through opioid dose usage was calculated as the product of prescribed dose per use, and the number of uses per day. If participants took more than 1 different break-through opioid for more than 1 day, the sum of morphine equivalents dose usages for each break-through opioid was calculated for the summary.
  Change in daily break-through opioid dose was calculated as: End of Treatment daily break-through opioid dose - Baseline daily break-through opioid dose.
  A negative value indicates a decrease in dose from Baseline.
Time Frame: Baseline, End of Treatment (Day 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg (morphine equivalent)
Arm/Group | Nabiximols | Placebo (GA-0034)
Number analyzed (Participants) | 199 | 198
mg (morphine equivalent) | 0.1 (22.2) | 1.8 (23.6)

11. Secondary Outcome: Change From Baseline In NRS Constipation At Last Visit (Up To Day 36)
Description: Participants indicated level of constipation on an 11-point NRS, where a score of 0 was "no constipation", and 10 was "constipation as bad as you can imagine." Last visit refers to the last visit that a participant completed the assessment; this could be either Day 22 or Day 36.
  Change in NRS constipation score was calculated as: Last Visit NRS constipation score - Baseline NRS constipation score.
  A negative value indicates improvement in condition from Baseline.
Time Frame: Baseline, Last Visit (up to Day 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nabiximols | Placebo (GA-0034)
Number analyzed (Participants) | 172 | 178
units on a scale | -0.6 (2.9) | -0.3 (2.8)

ADVERSE EVENTS:
Time Frame: Up to Day 43 post-randomization
Arm/Group | Nabiximols | Placebo (GA-0034)
Serious Adverse Events (participants affected / at risk) | 47/199 | 43/198
Other Adverse Events (participants affected / at risk) | 69/199 | 53/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nabiximols (N=199) | Placebo (GA-0034) (N=198)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 2
Mouth Haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Device Occlusion (General disorders) | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 1 | 2
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 31 | 28
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 1
Completed Suicide (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 1 | 0
Hallucination, Visual (Psychiatric disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nabiximols (N=199) | Placebo (GA-0034) (N=198)
Nausea (Gastrointestinal disorders) | 31 | 20
Dizziness (Nervous system disorders) | 16 | 8
Vomiting (Gastrointestinal disorders) | 15 | 11
Decreased Appetite (Metabolism and nutrition disorders) | 14 | 12
Constipation (Gastrointestinal disorders) | 11 | 13
Fatigue (General disorders) | 12 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days